CLINICAL TRIAL: NCT02456961
Title: Comparative Study of Results of Standard Corneal Collagen Crosslinking Versus Transepithelial Corneal Crosslinking by Iontophoresis of Riboflavin: a Randomized Control Trial
Brief Title: Standard Corneal Collagen Crosslinking Versus Transepithelial Corneal Crosslinking by Iontophoresis of Riboflavin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ufa Eye Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCXL-ionto
Record Dates: First submitted 2015-05-20; First posted 2015-05-29 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Keratoconus
Keywords: Collagen crosslinking (CXL); Standard corneal crosslinking (CXL); Transepithelial CXL; Iontophoresis; Riboflavin
MeSH Terms: conditions — Keratoconus | interventions — Corneal Cross-Linking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard epithelium-off CXL (Active Comparator): Removing the central 8-10mm of the epithelium and applying a riboflavin solution (0.1% riboflavin-5-phosphate and 20% dextran T-500) to the corneal surface 30 minutes before irradiation and at 5 minutes intervals during the course of a 30 minute exposure to 370 nm UVA with an irradiance of 3 mWcm-2 (UFalink, Russian Federation)
  Interventions: Procedure: epithelium-off; Procedure: Corneal collagen crosslinking; Drug: Dextralink; Device: UFalink
- Transepithelial CXL via iontophoresis of riboflavin (Experimental): impregnation of the cornea with a riboflavin 0.1% hypotonic solution is performed by using an iontophoresis device (galvanizator; Potok-1, Russian Federation). The passive electrode (anode) was applied to the inferior part of the cervical vertebrae. The active electrode (cathode), a bath tube (glass or plastic - 10-12 ml) is applied to the open eye,then r the tube is taped to the skin of the orbital margins and filled with riboflavin 0.1%. The current intensity is initially 0.2 mA and then gradually increased to 1.0 mA at 0.2 mA for 1 minute at 10-second intervals increments to determine individual tolerance. The total time that the riboflavin administration is 10 minutes.
  Standard surface UVA irradiation (370 nm, 3 mW/cm2) using UFalink device, (Russian Federation) is then applied at a 5-cm distance for 30 minutes with continuing hypotonic riboflavin drops every 2 minutes
  Interventions: Procedure: iontophoresis of riboflavin; Procedure: Corneal collagen crosslinking; Device: galvanizator, Potok-1; Drug: Riboflavin 0,1%; Device: UFalink

INTERVENTIONS:
Procedure: iontophoresis of riboflavin
  Arms: Transepithelial CXL via iontophoresis of riboflavin
Procedure: epithelium-off
  Arms: Standard epithelium-off CXL
Procedure: Corneal collagen crosslinking — Standard surface UVA irradiation (370 nm, 3 mW/cm2; UFalink, Russian Federation) was then applied at a 5-cm distance for 30 minutes. During UVA exposure, hypotonic riboflavin drops were continued every 2 minutes.
Device: galvanizator, Potok-1 — Device for providing iontophoresis procedure
  Arms: Transepithelial CXL via iontophoresis of riboflavin
Drug: Dextralink — Riboflavin 0,1% + Dextran T-500
  Arms: Standard epithelium-off CXL
Drug: Riboflavin 0,1%
  Arms: Transepithelial CXL via iontophoresis of riboflavin
Device: UFalink — device for UVA irradiation - providing UVA light - 370 nm, 3 mW/cm2

SUMMARY:
The standard CXL technique involves removal of the epithelium to enable riboflavin to penetrate into stromal tissue, to avoid epithelial debridement and increasing the patient's comfort and safety transepithelial corneal crosslinking (CXL) was suggested. Iontophoresis of riboflavin is one of approach for riboflavin impregnation.

In this study, the investigators compared the results of standard corneal crosslinking (CXL) and transepithelial CXL via iontophoresis of riboflavin after 24 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* Documented progressive KC (by Pentacam and/or corneal topography imaging).
* A clear central cornea.
* A minimal corneal thickness of ≥ 400 µm at the thinnest corneal location (Pentacam imaging).
* Minimal Snellen corrected distance visual acuity of ≥ 0.4.
* Patient age of ≥ 18 years.

Exclusion Criteria:

* Corneal scarring.
* History of epithelial healing problems.
* History or presence of ocular infection (such as herpes keratitis)
* Pregnancy and/or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2010-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Kmax, D | 2 years
  Using topography measurements, clinical stabilisation is defined as an increase of no more than 1 diopter of the maximum keratometry value over the preoperative maximum keratometry value

SECONDARY OUTCOMES:
Corneal thickness, μm, as measured by OCT tomography | 2 years
  Using optical coherence tomography to estimate the pachymetry changes
Visual acuity as assessed by Decimal system | 2 years
  Decimal visual acuity assessed on a study later was converted to the logarithm of minimal angle of resolution (logMAR).

CONTACTS AND LOCATIONS:
Overall Officials: Mukharram Bikbov, Professor, Study Chair — Ufa Eye Research Institute